CLINICAL TRIAL: NCT04933461
Title: Simulated Clinical Use Testing to Evaluate Sharps Injury Prevention Features of HTL-STREFA's Safety Lancets (Test C)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HTL-Strefa S.A. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Test C
Record Dates: First submitted 2021-06-09; First posted 2021-06-21 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Accident Injury
Keywords: safety lancet; capillary blood sampling; accidental needle-stick injury
MeSH Terms: conditions — Accidental Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simulation of skin pricking by using Medlance Plus (Other): Estimation of the true failure rate of the device. Estimation of the sharps' injury prevention feature of the tested safety lancets are effective in preventing needle stick injuries.
  Interventions: Device: Safety lancet
- Simulation of skin pricking by using myLance (Other): Estimation of the true failure rate of the device. Estimation of the sharps' injury prevention feature of the tested safety lancets are effective in preventing needle stick injuries.
  Interventions: Device: Safety lancet

INTERVENTIONS:
Device: Safety lancet — There are sterile, single-use safety lancets designed for the sampling of capillary blood from the fingertip of patients.

SUMMARY:
A simulated clinical use testing to evaluate the Medlance Plus and myLance sharps injury prevention feature in accordance with the FDA's guidance on medical devices with sharps injury prevention features.

DETAILED DESCRIPTION:
This study aims to evaluate the safety of the use of the following safety lancets: Medlance Plus and myLance in the prevention of needle-stick injury (NSI) and to evaluate the user's opinion with regard to the handling characteristics of the medical devices.

The simulated use clinical study involves healthcare professionals (HCPs) who routinely use safety lancets to collect blood samples.

ELIGIBILITY:
Inclusion Criteria:

* evaluators who routinely use safety lancets to collect capillary blood samples (prevention of the learning curve artifacts)
* evaluators will be United States (US) residents
* evaluators can read, write, and speak English
* evaluators are at least 18 years old
* evaluators are able to understand and provide signed consent for the study
* evaluators are willing to comply with the study protocol, including being willing to answer questions and complete questionnaires.
* evaluators have no concerns about the ability to perform the simulated skin pricking.

Exclusion Criteria:

* evaluators who do not routinely use safety lancets to collect capillary blood samples,
* evaluators who cannot read, write, and speak English,
* evaluators or a family member have a business or consulting relationship with a pharmaceutical or medical device company, or
* evaluators who have participated in a product evaluation or marketing study involving safety lancets within the last six months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-09-24 (Actual); Primary Completion 2019-09-24 (Actual); Study Completion 2019-09-27 (Actual)

PRIMARY OUTCOMES:
The true failure rate of the tested devices. | At time of testing, up to 90 minutes
Effectiveness of the safety lancet's sharps injury prevention features. | At time of testing, up to 90 minutes
  Evaluator questionnaire using five-point response Likert scale (coded from 1 "strongly disagree" to 5 "strongly agree") to measure respondents' attitudes to a particular question or statement. Numbers assigned to Likert scale express a "greater than" relationship.

SECONDARY OUTCOMES:
Evaluation of the safety of the devices based on the evaluators' assessments. | At time of testing, up to 90 minutes ]
Evaluation of various aspects of the ease of use. | At time of testing, up to 90 minutes ]
Detection of any handling, usability questions / issues associated with the device. | At time of testing, up to 90 minutes ]

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Chicago office, Chicago, Illinois
  - Boston office, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No